CLINICAL TRIAL: NCT00337103
Title: A Phase III Open Label, Randomized Two-Parallel-Arm Multicenter Study of E7389 Versus Capecitabine in Patients With Locally Advanced or Metastatic Breast Cancer Previously Treated With Anthracyclines and Taxanes
Brief Title: E7389 Versus Capecitabine in Patients With Locally Advanced or Metastatic Breast Cancer Previously Treated With Anthracyclines and Taxanes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-301
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Eribulin Mesylate
- 2 (Active Comparator)
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Eribulin Mesylate — 1.4 mg/m^2 intravenous (IV) infusion given over 2-5 minutes on Days 1 and 8 every 21 days
  Arms: 1
Drug: Capecitabine — Capecitabine 2.5 g/m^2/day administered orally twice daily in two equal doses on Days 1 to 14 every 21 days
  Arms: 2

SUMMARY:
The purpose of this study is to compare E7389 versus capecitabine in patients with locally advanced or metastatic breast cancer who are refractory to the most recent chemotherapy. This is an open-label, randomized, two-parallel arm study. Patients will be randomized to receive either E7389 or capecitabine on a one-to-one ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically or cytologically confirmed carcinoma of the breast. Every effort should be made to ensure that paraffin embedded tissue or slides from the diagnostic biopsy or surgical specimen are available for confirmation of diagnosis.
2. Patients with locally advanced or metastatic disease who have received up to three prior chemotherapy regimens, and no more than two prior regimens for advanced and/or metastatic disease.

   * Regimens must have included an anthracycline (e.g., doxorubicin, epirubicin) and a taxane (e.g., paclitaxel, docetaxel), either in combination or in separate regimens.
   * Patients with known human epidermal growth factor 2 (HER2/neu) over-expressing tumors may additionally have been treated with trastuzumab in centers where this treatment is available.
   * Patients with known estrogen and/or progesterone receptor-expressing tumors may have additionally been treated with hormonal therapy.
3. Resolution of all chemotherapy or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy <= Grade 2 and alopecia.
4. Age >= 18 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
6. Life expectancy of >= 3 months.
7. Adequate renal function as evidenced by serum creatinine <1.5 mg/dL or calculated creatinine clearance > 50 mL/minute (min) per the Cockcroft and Gault formula.
8. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) >= 1.5 x 10^9/L, hemoglobin >= 10.0 g/dL (a hemoglobin < 10.0 g/dL acceptable if it is corrected by growth factor or transfusion), and platelet count >= 100 x 10^9/L.
9. Adequate liver function as evidenced by bilirubin <= 1.5 times the upper limits of normal (ULN) and alkaline phosphatase, alanine transaminase (ALT), and aspartate transaminase (AST) <= 3 x ULN (in the case of liver metastases <= 5 x ULN), or in case of bone metastases, liver specific alkaline phosphatase <= 3 x ULN.
10. Patients willing and able to complete the EORTC (European Organization for Research on the Treatment of Cancer) quality of life questionnaire (QLQ-C30 with breast cancer module QLQ-BR23) and to record their pain level on the Visual Analog Scale (VAS).
11. Patients willing and able to comply with the study protocol for the duration of the study.
12. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion Criteria:

1. Patients who have received more than three prior chemotherapy regimens for their disease, including adjuvant therapies, or patients who have received more than two prior chemotherapy regimens for advanced disease (other therapies are allowed e.g., anti-estrogens, trastuzumab and radiotherapy).
2. Patients who have received capecitabine as a prior therapy for their disease.
3. Patients who have received chemotherapy, radiation, or biological therapy within two weeks, or hormonal therapy, within one week before study treatment start, or any investigational drug within four weeks before study treatment start.
4. Radiation therapy encompassing > 30% of marrow.
5. Prior treatment with mitomycin C or nitrosourea.
6. Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen.
7. Patients with brain or subdural metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment with study treatment. Any symptoms attributed to brain metastases must be stable for at least 4 weeks before starting study treatment; radiographic stability should be determined by comparing a contrast-enhanced Computed Tomography Scan (CT) or Magnetic Resonance Imaging (MRI) brain scan performed during screening to a prior scan performed at least 4 weeks earlier.
8. Patients with meningeal carcinomatosis.
9. Patients who are receiving anti-coagulant therapy with warfarin or related compounds, other than for line patency, and cannot be changed to heparin-based therapy, are not eligible. If a patient is to continue on mini-dose warfarin, then the prothrombin time (PT)/international normalized ratio (INR) must be closely monitored.
10. Women who are pregnant or breast-feeding; women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test; women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception (considered to be two methods of contraception, one of which must be a barrier method, e.g. condom, diaphragm or cervical cap). Perimenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
11. Severe/uncontrolled intercurrent illness/infection.
12. Significant cardiovascular impairment (history of congestive heart failure > New York Heart Association [NYHA] Grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia).
13. Patients with organ allografts requiring immunosuppression.
14. Patients with known positive human immunodeficiency virus (HIV) status.
15. Patients who have had a prior malignancy, other than carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated >= 5 years previously with no subsequent evidence of recurrence.
16. Patients with pre-existing neuropathy > Grade 2.
17. Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
18. Patients who participated in a prior E7389 clinical trial.
19. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1276 (Actual)
Dates: Start 2006-09-20 (Actual); Primary Completion 2012-03-12 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (167):
- United States (13):
  - Anaheim, California
  - La Verne, California
  - Poway, California
  - Centralia, Illinois
  - Augusta, Maine
  - Boston, Massachusetts
  - Jefferson City, Missouri
  - Lebanon, New Hampshire
  - Ephrata, Pennsylvania
  - Cookeville, Tennessee
  - Germantown, Tennessee
  - Amarillo, Texas
  - Wenatchee, Washington
- Argentina (13):
  - Hospital General de Agudos Teodoro Alvarez, Ciudad Autonoma, Buenos Aires
  - Instituto Argentino de Diagnostico y Tratamiento, Cuidad Autonoma de Buenos Aires, Buenos Aires
  - La Plata, Buenos Aires
  - Pilar, Buenos Aires
  - Corporacion Medica General San Martin, San Martín, Buenos Aires
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Bahía Blanca
  - Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Ciudad Autonoma
  - Mendoza
  - Santa Fe
- Australia (10):
  - Bankstown Hospital, Oncology Trials Unit, Bankstown, New South Wales
  - Hornsby, New South Wales
  - Liverpool Hospital, Cancer Therapy Centre, Liverpool, New South Wales
  - Ashford Cancer Centre, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Saint Vincent's Hospital, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Epworth Freemasons Hospital, East Melbourne
  - Sir Charles Gairdner Hospital, Dept. of Medical Oncology, Nedlands
  - Mater Adult Hospital, South Brisbane
- Belgium (4):
  - OLVZ Aalst, Oncology Service, Aalst
  - Institut Jules Bordet, Medical Oncology Unit, Brussels
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Centre Hosptialier Universitaire Sart Tilman Liege, Liège
- Brazil (15):
  - Florianópolis
  - Associacao Hospital de Caridade Ijui, Ijuí
  - Instituto de Oncologia Ltda, Jundiaí
  - Proonco Centro de Tratamento Oncologico, Londrina
  - Hospital de Clinicas de Porto Alegre, Servicio de Oncologia, Porto Alegre
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Servico de Quimioterapia de Pernambuco-SEQUIPE, Recife
  - Instituto Ribeiraopretano de Combate ao Cancer, Ribeirão Preto
  - Nucleo de Oncologia da Bahia, Salvador
  - Faculdade de Medicina do ABC, Santo André
  - Grupo Paulista de Oncologia Integrada Ltda, São Paulo
  - Hospital das Clinicas de Faculdade de Medicina da Universidade de Sao, São Paulo
  - Hospital do Cancer de Sao Paulo-AC Camargo, São Paulo
  - Hospital do Cancer de Sao Paulo-AC. Camargo, São Paulo
  - Instituto Brasileiro de Controle do Cancer-IBCC, São Paulo
- Bulgaria (9):
  - Burgas
  - Gabrovo
  - Pleven
  - Plovdiv
  - Rousse
  - Shumen
  - Sofia
  - Stara Zagora
  - Varna
- Canada (5):
  - Kingston, Ontario
  - Montreal General Hospital, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Montreal, Hopital Notre Dame, Montreal
  - Thunder Bay Regional Health Science Centre Northwestern Ontario, Thunder Bay
- Czechia (4):
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - Onkologicka Klinika, Fakutni Nemocnice, Olomouc
  - 1. LF UK, Ustav radiacnej onkologie, Prague
  - Krajska nemocnice T. Bati, Zlin Poiters
- France (3):
  - Centre Hospitalier La Roche sur Yon, CHD les Oudairies, La Roche-sur-Yon
  - CHU de Poitiers, Service d'Oncologie Medicale, Poitiers
  - Hopital Nord Saint-Etienne, Saint-Priest-en-Jarez
- Germany (5):
  - Augusta-Kranken-Anstalt, Klinik fur Hamatologie und Onkologie, Bochum
  - Hamburg
  - Homburg
  - Universitatsfrauenklinik Magdeburg, Magdeburg
  - Rostock
- Pátrai, Greece
- Hungary (7):
  - Gyor, Budapest
  - Debrecen University, Debrecen
  - Debrecen
  - Gyula
  - Pecsi Tudomanyegyetem, Onkoterapias Intezet, Pécs
  - Szeged
  - Veszprém
- Israel (7):
  - Barzilai Medical Center, Ashkelon
  - Soroka Medical Center, Beersheba
  - Sharet Institute of Oncology, Jerusalem
  - Meir Hospital, Sapir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (8):
  - Ancona
  - Unita Operativa de Oncologia, Lugo
  - Meldola
  - Modena
  - Azienda Ospedaliera San Salvatore, Pesaro
  - Ospedale Civile S. Maria delle Croci, Ravenna
  - UO di Onco-ematologia, Rimini
  - Sassari
- Mexico (3):
  - Centro Estatal de Cancerologia, Chihuahua City
  - Monterrey
  - Consultorio del Dr. Trigueros, Morelia
- Poland (9):
  - Regionalny Osrodek Onkologii, Bialystok
  - Bytom
  - Elblag
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Krakow
  - Olsztyn
  - Rybnik
  - Torun
  - Wojewodzki Szpital Specjalistyczny, Wroclaw
- Romania (7):
  - Cluj-Napoca, Cluj
  - Spitalul Militar Central Bucuresti, Bucharest
  - Bucharest
  - Cluj-Napoca
  - Centrul de Oncologie Medicala, Iași
  - Spitalul Clinic Judetean Sibiu, Sibiu
  - Timișoara
- Russia (15):
  - Regional Oncology Dispensary, Yaroslavl, Yaroslavlr
  - Barnaul
  - Kazan'
  - Kirov
  - Krasnodar
  - Blokhin Cancer Research Centre, Moscow
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Sochi
  - Tomsk
  - Vladimir
- Singapore, Singapore
- South Africa (7):
  - Mayville, Durban
  - Pretoria, Gaunteng
  - Groenkloof, Pretoria
  - Panorama Medical Centre, Cape Town
  - Durban
  - Johannesburg
  - Sandton
- Spain (6):
  - Barakaldo, Vizcaya
  - A Coruña
  - Barcelona
  - Guadalajara
  - Seville
  - Valencia
- Taiwan (5):
  - Changhua
  - Taichung
  - Tainan
  - Taipei
  - Yung-Kang City
- Ukraine (10):
  - Chernihiv
  - Dnipro
  - Donetsk
  - Kharkiv
  - Khmelnytskyi
  - Kiev
  - Kryvyi Rih
  - Kyiv
  - Lviv
  - Odesa

REFERENCES:
- [Derived] Twelves C, Awada A, Cortes J, Yelle L, Velikova G, Olivo MS, Song J, Dutcus CE, Kaufman PA. Subgroup Analyses from a Phase 3, Open-Label, Randomized Study of Eribulin Mesylate Versus Capecitabine in Pretreated Patients with Advanced or Metastatic Breast Cancer. Breast Cancer (Auckl). 2016 Jun 28;10:77-84. doi: 10.4137/BCBCR.S39615. eCollection 2016. PMID 27398025
- [Derived] Twelves C, Cortes J, Kaufman PA, Yelle L, Awada A, Binder TA, Olivo M, Song J, O'Shaughnessy JA, Jove M, Perez EA. "New" metastases are associated with a poorer prognosis than growth of pre-existing metastases in patients with metastatic breast cancer treated with chemotherapy. Breast Cancer Res. 2015 Dec 9;17(1):150. doi: 10.1186/s13058-015-0657-1. PMID 27391598
- [Derived] Cortes J, Hudgens S, Twelves C, Perez EA, Awada A, Yelle L, McCutcheon S, Kaufman PA, Forsythe A, Velikova G. Health-related quality of life in patients with locally advanced or metastatic breast cancer treated with eribulin mesylate or capecitabine in an open-label randomized phase 3 trial. Breast Cancer Res Treat. 2015 Dec;154(3):509-20. doi: 10.1007/s10549-015-3633-7. Epub 2015 Nov 14. PMID 26567010
- [Derived] Kaufman PA, Awada A, Twelves C, Yelle L, Perez EA, Velikova G, Olivo MS, He Y, Dutcus CE, Cortes J. Phase III open-label randomized study of eribulin mesylate versus capecitabine in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2015 Feb 20;33(6):594-601. doi: 10.1200/JCO.2013.52.4892. Epub 2015 Jan 20. PMID 25605862
- [Derived] Twelves C, Cortes J, Vahdat LT, Wanders J, Akerele C, Kaufman PA. Phase III trials of eribulin mesylate (E7389) in extensively pretreated patients with locally recurrent or metastatic breast cancer. Clin Breast Cancer. 2010 Apr;10(2):160-3. doi: 10.3816/CBC.2010.n.023. PMID 20299316

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1276 participants were enrolled and screened, of which 174 were screen failures and 1102 were randomized in the study. Of the randomized participants, 1090 participants received the study treatment.
Groups:
- Eribulin Mesylate 1.4 mg/m^2: Eribulin mesylate 1.4 milligram per meter square (mg/m^2) intravenous (IV) infusion given over 2-5 minutes on Days 1 and 8 every 21 days.
- Capecitabine 2.5 g/m^2/Day: Capecitabine : Capecitabine 2.5 gram per meter square per day (g/m^2/day) administered orally twice daily in two equal doses on Days 1 to 14 every 21 days.
Period: Overall Study
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Started | 554 | 548
Treated (Safety Population) | 544 | 546
Completed | 0 | 0
Not Completed | 554 | 548
Not completed — Progressive Disease | 414 | 410
Not completed — Adverse Event | 45 | 59
Not completed — Subject Choice | 34 | 27
Not completed — Clinical Progression | 27 | 24
Not completed — Physician Decision | 15 | 14
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Other | 5 | 6
Not completed — Entry Criteria Not Met | 4 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Eribulin Mesylate 1.4 mg/m^2: Eribulin mesylate 1.4 mg/m^2 intravenous (IV) infusion given over 2-5 minutes on Days 1 and 8 every 21 days.
- Capecitabine 2.5 g/m^2/Day: Capecitabine : Capecitabine 2.5 g/m^2/day administered orally twice daily in two equal doses on Days 1 to 14 every 21 days.
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day | Total
Number analyzed (Participants) | 554 | 548 | 1102
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (10.37) | 52.8 (10.20) | 53.3 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 554 | 548 | 1102
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 18 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 16 | 31
  White | 496 | 495 | 991
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was measured from the date of randomization until the date of death from any cause, or the last date the participant was known to be alive. Participants who were lost to follow-up or who were alive at the date of data cutoff were censored. The censoring rules for OS were as follows: 1) if the participant was still alive at data cutoff, the date of data cutoff was considered the end date, and 2) if the participant was lost to follow-up before data cutoff, the date they were last known to be alive was considered the end date. Participants who survived past the end of the study were counted as in the full study period. If death occurred after data cutoff, the end date was to be censored at the time of data cutoff.
Time Frame: From date of randomization until date of death from any cause, assessed up to data cutoff date of 12 Mar 2012, or up to approximately 6 years
Population: Data was analyzed using the Intent-to-Treat (ITT) Population defined as all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 554 | 548
days | 484 [462 to 536] | 440 [400 to 487]

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time (in days) from the date of randomization to the date of the first sign of disease progression based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 (v 1.1) or date of death, regardless of cause. Disease progression was measured by computed tomography (CT) and magnetic resonance imaging (MRI) performed on lesions targeted at baseline for tumor assessment. Disease progression (as assessed by independent review of the imaging scans) per RECIST v 1.1 was defined as at least a 20% increase in the sum of the diameters of the target lesions (taking as reference the smallest sum on study, including the baseline sum if that is the smallest), and an absolute increase of at least 5 millimeter (mm). Note that the appearance of one or more new lesions was also considered as disease progression.
Time Frame: From date of randomization to the date of disease progression or death (whichever occurred first), assessed up to data cutoff date of 12 Mar 2012 or up to approximately 6 years
Population: Data was analyzed using the ITT Population defined as all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 554 | 548
Days | 126 [106 to 131] | 129 [120 to 147]

3. Secondary Outcome: Change From Baseline in Global Health Status/Quality of Life (QoL) Measured by European Organization for the Treatment of Cancer Quality of Life Core Questionnaire Scores Based on Core 30 Items (EORTC-QLQ-C30) at Week 6
Description: EORTC-QLQ-C30:cancer-specific instrument with 30 questions to assess the participant QoL. First 28 questions used to evaluate 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, nausea and vomiting, pain) and other single items(dyspnoea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Each of these 28 questions assessed on 4-point scale(1=not at all, 2=a little, 3=quite a bit, 4=very much); functional scales: higher score=better level of functioning; symptom scale: higher score=more severe symptoms; for single items: higher score= more severe problem. Last 2 questions used to evaluate global health status (GHS)/QoL. Each question was assessed on 7-point scale (1=very poor to 7=excellent). Scores averaged, transformed to 0-100 scale; higher score=better quality of life/better level of functioning.
Time Frame: Baseline and Week 6
Population: Data was analyzed using the ITT Population defined as all participants who were randomized. Here,"overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 438 | 406
units on a scale | 0.1 (19.23) | 1.7 (20.69)

4. Secondary Outcome: Change From Baseline in European Organization for the Treatment of Cancer Quality of Life Core Questionnaire Scores Based on Breast Cancer Specific 23 Items (EORTC-QLQ- BR 23) at Week 6
Description: EORTC-QLQ-BR23:disease-specific module for breast cancer developed as a supplement for the EORTC-QLQ-C30 to assess quality of life of participants with breast cancer. The scores from 23 items of QLQ-BR23 included functional scales (body image, sexual functioning, sexual enjoyment, future perspective), symptom scales (systemic therapy side effects, breast symptoms, arm symptoms, upset by hair loss). Each item was rated on a scale of 1 to 4 to record level of intensity (1= not at all, 2= a little, 3= quite a bit, 4= very much) within each scales. Scores averaged and transformed to 0-100 scale. High score indicated high/better level of functioning/healthy functioning. Negative change from Baseline indicated deterioration in QOL and positive change from Baseline indicated an improvement in QOL.
Time Frame: Baseline and Week 6
Population: Data was analyzed using the ITT Population defined as all participants who were randomized. Here,"number analyzed" signifies the participants who were evaluable for this outcome measure for individual row.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 554 | 548
units on a scale
  Body Image: number analyzed (Participants) | 441 | 411
  Body Image | 0.7 (21.26) | 4.8 (21.80)
  Sexual functioning: number analyzed (Participants) | 418 | 381
  Sexual functioning | 1.2 (14.75) | -0.1 (16.62)
  Sexual enjoyment: number analyzed (Participants) | 82 | 96
  Sexual enjoyment | 0.8 (21.58) | 3.1 (17.49)
  Future perspective: number analyzed (Participants) | 439 | 410
  Future perspective | 7.7 (28.48) | 10.0 (30.84)
  Systemic therapy side effects: number analyzed (Participants) | 440 | 415
  Systemic therapy side effects | 4.5 (15.55) | -1.2 (14.73)
  Breast Symptoms: number analyzed (Participants) | 434 | 407
  Breast Symptoms | -3.4 (16.55) | -3.6 (16.20)
  Arm Symptoms: number analyzed (Participants) | 437 | 411
  Arm Symptoms | -4.2 (17.94) | -3.4 (18.65)
  Upset by hair loss: number analyzed (Participants) | 91 | 56
  Upset by hair loss | -4.4 (32.66) | -10.1 (29.76)

5. Secondary Outcome: Objective Response Rate (ORR): Independent Review
Description: ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v 1.1). CR is defined as disappearance of all target legions and non-target lesions. All pathological lymph nodes (whether target and non-target), must have reduction in their short axis to less than 10 mm. PR is defined as at least 30% decrease in the sum of the long diameter LD (hereafter referred to as sum of LD) of all target lesions, as compared with Baseline summed LD.
Time Frame: From date of randomization until date of first documentation of CR or PR, assessed up to data cutoff date of 12 Mar 2012 or up to approximately 6 years
Population: Data was analyzed using the ITT Population defined as all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 554 | 548
percentage of participants | 11.0 [8.5 to 13.9] | 11.5 [8.9 to 14.5]

6. Secondary Outcome: Duration of Response (DOR): Independent Review
Description: DOR was defined as the time from first documented CR or PR until disease progression or death from any cause for those participants with a confirmed PR or CR measured by RECIST v1.1. CR defined as disappearance of all target and non-target lesions. All pathological lymph nodes(whether target and non-target), must have reduction in their short axis to less than 10 mm. PR defined as at least 30% decrease in the sum of the long diameter LD (hereafter referred to as sum of LD) of all target lesions, as compared with Baseline summed LD.
Time Frame: From first documented CR or PR until date of recurrent or progressive disease or death, assessed up to data cutoff of date of 12 Mar 2012 or up to approximately 6 years
Population: Data was analyzed using for a subset of participants in the ITT Population who had a response. Here, "overall number of participants analyzed" are the participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 61 | 63
days | 198 [150 to 273] | 330 [208 to 541]

7. Secondary Outcome: Overall Survival Rate
Description: One-, two-, and three- year's survival rates were defined as the percentage of participants who were alive at one, two, and three years respectively, and estimated using the Kaplan-Meier method and Greenwood Formula.
Time Frame: From the date of randomization to Year 1, 2 and 3
Population: Data was analyzed using the ITT Population defined as all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 554 | 548
percentage of participants
  At 1-year | 0.644 [0.604 to 0.684] | 0.580 [0.538 to 0.622]
  At 2-years | 0.328 [0.289 to 0.368] | 0.298 [0.259 to 0.337]
  At 3-years | 0.178 [0.144 to 0.212] | 0.145 [0.113 to 0.177]

8. Secondary Outcome: Change From Baseline in Pain Intensity by Visual Analog Scale (VAS) Until 30 Days After the Last Dose of Study Drug
Description: Pain intensity was measured by marking a single vertical line that crosses a 1-100 mm unmarked VAS scale. The left-end of the visual analog scale was labelled "least possible pain" and the right-end of the visual analog scale was labelled "worst possible pain". The pain rating ranged from 0 to 100, with a higher score indicating more pain. A negative change score indicated improvement.
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (up to approximately 6 years 3 months)
Population: Data was analyzed using the ITT Population defined as all participants who were randomized. Here, "overall number of participants analyzed" are the participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 431 | 431
units on a scale | -3.7 (22.80) | 0.4 (22.90)

9. Secondary Outcome: Number of Participants With Consumption of Analgesics During the Study
Description: Participants took analgesics as concomitant pain medications which are defined as pain medications that (1) started before the first dose of study drug and were continuing at the time of the first dose of study drug, or (2) started on/after the day of the first dose of study drug up to 30 days after the last dose of study drug medication
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (up to approximately 6 years 3 months)
Population: Data was analyzed using safety population defined as all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 544 | 546
Participants | 222 | 196

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAEs included both SAEs as well as non-SAEs.
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (up to approximately 6 years 3 months)
Population: Data was analyzed using safety population defined as all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 544 | 546
Participants
  TEAEs | 512 | 494
  SAEs | 95 | 115

11. Secondary Outcome: Number of Participants With Treatment-emergent Markedly Abnormal Laboratory Parameter Values
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (up to approximately 6 years 3 months)
Population: Data was analyzed using safety population defined as all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 544 | 546
Participants | 362 | 224

12. Secondary Outcome: Number of Participants Who Took at Least One Concomitant Medication
Description: Concomitant medications included medications that either (1) started before the first dose of study drug and were continuing at the time of the first dose of study drug, or (2) started on or after the first dose of study drug up to 30 days after the last dose of study drug.
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (up to approximately 6 years 3 months)
Population: Data was analyzed using safety population defined as all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 544 | 546
Participants | 496 | 483

13. Secondary Outcome: Duration of Eribulin Mesylate Exposure
Description: Data have been reported per primary analysis completion stage and final analysis completion stage. After primary analysis completion (at cutoff date of 12 March 2012), only 10 participants were still receiving study treatment.
Time Frame: Up to approximately 6 years for primary analysis completion stage, Up to approximately 6 years 2 months for final analysis completion stage
Population: Data was analyzed using safety population defined as all participants who received at least one dose of study treatment. Here, "number analyzed" signifies the participants who were evaluable at individual stage for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
Number analyzed (Participants) | 544 | 546
days
  At primary analysis completion stage | 125.0 [21 to 1372] | 119.0 [21 to 1442]
  At final analysis completion stage: number analyzed (Participants) | 5 | 5
  At final analysis completion stage | 1743.0 [1561 to 2219] | 1506.0 [1175 to 2296]

14. Secondary Outcome: Plasma Concentrations of Eribulin Mesylate
Time Frame: Cycle 1 Day 1: 5-10 minutes(min), 15-30 min, 30-60 min, 60-90 min, 2-4 hours(hrs), 4-8 hrs, 10-24 hrs, 48-72 hrs, 72-96 hrs, 96-120 hrs after the start of infusion of Eribulin mesylate (Duration of each cycle is 21 days)
Population: Pharmacokinetic (PK) analysis set included all participants who have received at least one dose of E7389 and have at least one quantifiable E7389 concentration. Here, "number analyzed" signifies the participants who were evaluable for this outcome measure for given time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Eribulin Mesylate 1.4 mg/m^2
Number analyzed (Participants) | 173
nanogram per milliliter (ng/mL)
  5-10 minutes: number analyzed (Participants) | 172
  5-10 minutes | 415.8 (719.5)
  15-30 minutes: number analyzed (Participants) | 57
  15-30 minutes | 152.6 (70.51)
  30-60 minutes: number analyzed (Participants) | 58
  30-60 minutes | 95.5 (87.90)
  60-90 minutes: number analyzed (Participants) | 58
  60-90 minutes | 52.7 (79.33)
  2-4 hours: number analyzed (Participants) | 85
  2-4 hours | 20.7 (32.81)
  4-8 hours: number analyzed (Participants) | 78
  4-8 hours | 10.0 (5.40)
  10-24 hours: number analyzed (Participants) | 44
  10-24 hours | 5.8 (3.72)
  48-72 hours: number analyzed (Participants) | 40
  48-72 hours | 3.7 (2.58)
  72-96 hours: number analyzed (Participants) | 37
  72-96 hours | 2.4 (1.60)
  96-120 hours: number analyzed (Participants) | 41
  96-120 hours | 7.6 (38.75)

ADVERSE EVENTS:
Time Frame: First dose of study drug (Baseline) up to 30 days after last dose of study drug (up to approximately 6 years 3 months)
Description: Data was analyzed using Safety Population defined as all participants who received at least one dose of study treatment.
Arm/Group | Eribulin Mesylate 1.4 mg/m^2 | Capecitabine 2.5 g/m^2/Day
All-Cause Mortality (participants affected / at risk) | 442/544 | 459/546
Serious Adverse Events (participants affected / at risk) | 95/544 | 115/546
Other Adverse Events (participants affected / at risk) | 509/544 | 489/546
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2 (N=544) | Capecitabine 2.5 g/m^2/Day (N=546)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 17
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 10 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 4
Leukopenia (Blood and lymphatic system disorders) | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 5
Asthenia (General disorders) | 3 | 4
Fatigue (General disorders) | 3 | 4
Death (General disorders) | 2 | 2
General Physical Health Deterioration (General disorders) | 2 | 3
Multi-Organ Failure (General disorders) | 1 | 2
Extravasation (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 2
Generalized Edema (General disorders) | 0 | 1
Injection Site Extravasation (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 4
Cerebrovascular Accident (Nervous system disorders) | 2 | 2
Spinal Cord Compression (Nervous system disorders) | 2 | 2
Convulsion (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0
Facial Paresis (Nervous system disorders) | 1 | 0
Myoclonic Epilepsy (Nervous system disorders) | 1 | 0
Partial Seizures (Nervous system disorders) | 1 | 0
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1
Cerebellar Infarction (Nervous system disorders) | 0 | 1
Coma Hepatic (Nervous system disorders) | 0 | 1
Dysgeuesia (Nervous system disorders) | 0 | 1
Intracranial Pressure Increased (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Simple Partial Seizures (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4
Sepsis (Infections and infestations) | 2 | 4
Bronchopneumonia (Infections and infestations) | 1 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Pneumonia Klebsiella (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 0 | 2
Staphylococcal Infection (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oncologic Complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 9
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 15
Nausea (Gastrointestinal disorders) | 1 | 7
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1
Pericardial Effusion (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory Arrest (Cardiac disorders) | 0 | 1
Cardiogenic Shock (Cardiac disorders) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 2
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 2 | 3
Hypotension (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Shock Haemorrhagic (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Haemoglobin Decreased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Troponin Increased (Investigations) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Palmar-Plantar Erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 0 | 2
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Malignant Breast Lump Removal (Surgical and medical procedures) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2 (N=544) | Capecitabine 2.5 g/m^2/Day (N=546)
Neutropenia (Blood and lymphatic system disorders) | 292 | 87
Leukopenia (Blood and lymphatic system disorders) | 171 | 57
Anaemia (Blood and lymphatic system disorders) | 102 | 96
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 29
Fatigue (General disorders) | 91 | 82
Asthenia (General disorders) | 83 | 79
Pyrexia (General disorders) | 67 | 27
Oedema Peripheral (General disorders) | 35 | 36
Mucosal Inflammation (General disorders) | 26 | 35
Nausea (Gastrointestinal disorders) | 121 | 131
Diarrhoea (Gastrointestinal disorders) | 77 | 154
Vomiting (Gastrointestinal disorders) | 63 | 89
Constipation (Gastrointestinal disorders) | 42 | 46
Abdominal Pain (Gastrointestinal disorders) | 32 | 46
Abdominal Pain Upper (Gastrointestinal disorders) | 31 | 39
Stomatitis (Gastrointestinal disorders) | 27 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 188 | 22
Peripheral Sensory Neuropathy (Nervous system disorders) | 73 | 38
Headache (Nervous system disorders) | 67 | 55
Dizziness (Nervous system disorders) | 30 | 29
Back Pain (Musculoskeletal and connective tissue disorders) | 55 | 43
Bone Pain (Musculoskeletal and connective tissue disorders) | 50 | 42
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 47 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 30 | 8
Urinary Tract Infection (Infections and infestations) | 29 | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 49 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 44
Decreased Appetite (Metabolism and nutrition disorders) | 68 | 80
Alanine Aminotransferase Increased (Investigations) | 47 | 23
Aspartate Aminotransferase Increased (Investigations) | 43 | 27
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 | 22
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 | 38
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 244

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No